CLINICAL TRIAL: NCT06362616
Title: Preoperative Accelerated Partial Breast Irradiation in Patients With Locally Recurrent or Second Primary Breast Cancer
Acronym: PAPBI-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Medical Center Haaglanden (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N23PBD
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Recurrent breast cancer; Preoperative; Partial breast irradiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative accelerated partial breast re-irradiation (Experimental): Patients receive preoperative accelerated partial breast irradiation of the in situ tumor in the breast followed by repeat breast conserving surgery
  Interventions: Radiation: Preoperative accelerated partial breast irradiation; Procedure: Breast conserving surgery; Procedure: Sentinel node procedure; Procedure: Biopsy track removal

INTERVENTIONS:
Radiation: Preoperative accelerated partial breast irradiation — Patients will be treated with 5 x 5.2 Gray (Gy) preoperative accelerated partial breast irradiation of the in situ tumor in the breast
Procedure: Breast conserving surgery — Patients will be treated with breast conserving surgery.
Procedure: Sentinel node procedure — Patients will undergo a (repeat) sentinel node procedure.
Procedure: Biopsy track removal — The biopsy track will be surgically removed.

SUMMARY:
This study evaluates the acute toxicity and feasibility of repeat breast conserving therapy with preoperative accelerated partial breast re-irradiation (PAPBI) in female patients aged 51 years or older with ipsilateral recurrent or second primary low-risk breast cancer or DCIS.

DETAILED DESCRIPTION:
Standard treatment for an ipsilateral breast recurrence is a salvage mastectomy. However, repeat breast conserving therapy, involving breast conserving surgery (BCS) and postoperative re-irradiation, is a feasible alternative for a selected group of patients. In the primary setting, accelerated partial breast irradiation (APBI) is an international accepted treatment for a subset of breast cancer patients. Preoperative APBI (PAPBI) leads to low complication rates, limited fibrosis/induration in a small volume and good to excellent cosmetic results compared with results reported after postoperative APBI.

The aim of this study is to asses the acute toxicity and feasibility of repeat breast conserving therapy with PAPBI followed by BCS in patients aged 51 years or older with ipsilateral recurrent or second primary low-risk breast cancer or DCIS.

Patients undergo PAPBI 5 times (5 x 5.2 Gray). One-two weeks after completion of PAPBI, patients undergo BCS.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 51 years
* Ipsilateral breast cancer; recurrence or second primary
* Either histologically proven invasive adenocarcinoma (invasive adenocarcinoma with DCIS component is also accepted) or DCIS alone (calcification associated on imaging)
* Histologically proven estrogen receptor positive
* HER2neu negative
* In case of invasive adenocarcinoma: tumor size ≤ 3 cm. In case of DCIS alone: affected area ≤ 2.5 cm
* Grade I or grade II (biopsy)
* cN0M0 (No evidence of nodal or distant metastases on axillary ultrasound and, if indicated, positron emission tomography-computed tomography (PET-CT) scan)
* Unifocal lesions on mammogram and MRI (small satellite lesions adjacent to the tumor are accepted as long as it is suitable for local excision)
* Interval since completion of local treatment of primary tumor > 12 months
* Previous radiotherapy (whole breast or partial) of the ipsilateral breast
* Repeat breast conserving surgery feasible
* World Health Organization (WHO) performance ≤ 2
* Written informed consent
* The patient is legally competent

Exclusion Criteria:

* ≥ grade 3 radiotherapy toxicity in the breast after treatment of the primary tumor
* Previous boost radiotherapy is not allowed, UNLESS the protocol tumor lies outside of the original boost area
* Distant metastases and/or synchronous contralateral invasive or in situ carcinoma
* Invasive lobular carcinoma (ILC) or pleiomorphic lobular carcinoma in situ (LCIS)
* ER negative subtype
* Lymphovascular invasion in biopsy
* Neoadjuvant systemic treatment for the protocol tumor (except for pre-surgery hormonal therapy ≤ 2 months)
* (Planned) oncoplastic surgery with major tissue displacement
* Participation in another clinical trial that interferes with the locoregional treatment of this protocol.
* It is expected that dosimetric constraints cannot be met, such as lung/heart constraints.
* Patients with proven BRCA-mutations

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who were born as female
Enrollment: 31 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-10-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Acute post-treatment toxicity | 3,5 months
  Acute post-treatment toxicity from start of local treatment up to 3 months after end of local treatment, assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Values range form 0 to 5, with 5 being the worst value. At least grade ≥ 2 toxicity is scored as an event.

SECONDARY OUTCOMES:
Fibrosis/induration | 3 months
  Assessment of fibrosis/induration grade at 3 months after end of local treatment, assessed the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Values range form 0 to 5, with 5 being the worst value.
Patient-reported Outcome Measures (PROMS): EORTC Quality of Life Questionnaire (QLQ)-C30 | 3,5 months
  PROMs will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
Patient-reported Outcome Measures (PROMS): EORTC QLQ-BR23 | 3,5 months
  PROMs will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-BR23 questionnaire. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
Patient-reported Outcome Measures (PROMS): Patient's Questionnaire Cosmesis | 3,5 months
  PROMs will be assessed using the Patient's Questionnaire Cosmesis, adapted from Sneeuw et al. (1992). Patients score their cosmetic outcome by the following outcomes: very satisfied, satisfied, neutral, unsatisfied and very unsatisfied.
Cosmetic outcome according to the BCCT.core software program | 3,5 months
  Cosmetic outcome according to the Breast Cancer Conservative Treatment cosmetic results (BCCT.core) software program. The program returns an overall cosmetic outcome score (excellent, good, fair, or poor) based on the symmetry of the breasts, skin color, and scar visibility.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Scholten, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands